CLINICAL TRIAL: NCT02446951
Title: Implementation of a Clinical Decision Rule for Treatment of Neonatal Jaundice in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1404-061
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED Jaundice Patients: Patients presenting to the ED in either the implementation period or pre-implementation period.

SUMMARY:
Jaundice is a condition caused by elevated levels of bilirubin in the body otherwise known as hyperbilirubinemia. It occurs when there is an increase in bilirubin production or normal production with problems eliminating it from the body. Serum levels of bilirubin in excess of 5 mg/dL signifies clinical jaundice, yet more than half of full term infants experience these levels within the first week of life. For those patients who have markedly elevated serum bilirubin levels, which phototherapy cannot sufficiently treat, the use of exchange transfusions is a viable option within the hospital setting. In comparison, bili-blankets have been used as a form of phototherapy for those patients being treated in a home-based setting to reduce the likelihood of hospital readmissions.

DETAILED DESCRIPTION:
Background The rate of hospital admissions for hyperbilirubinemia (jaundice) has increased over the past 10 years. Jaundice is a condition caused by elevated serum levels of bilirubin due to an increase in bilirubin production or normal production with problems eliminating it from the body. Serum levels of bilirubin in excess of 5 mg/dL signify clinical jaundice; more than half of full term infants experience these levels within the first week of life.1 It is important for health care providers to distinguish infants experiencing physiologic jaundice as part of otherwise healthy development from those experiencing pathologic jaundice which, if not treated aggressively, can lead to irreversible damage of the central nervous system.2 Since 2000 there has been a 160% increase in the number of children readmitted to hospitals for jaundice after discharge from the hospital nursery.2 This dramatic increase is believed to be associated with the change in birth hospital culture as newborns are now typically discharged 48 hours after delivery while bilirubin levels are still on the rise. Bilirubin levels typically peak between the third and fifth day of life.3 The change in hospital discharge procedures results in circumstances where parents may present for medical care in an ED when their newborn starts to show symptoms of jaundice. This trend has been observed despite the implementation of routine bilirubin screening in many newborn nurseries. Similar to national trends, at Children's there has been a substantial increase in ED evaluations for jaundice; in 2012, 274 neonates younger than 7 days old were treated for jaundice in Children's EDs. Families may seek care in the ED as they may not have an established relationship with a Pediatrician or they may believe that their child requires an intervention that was only available in the ED setting. While some of these patients are ultimately admitted to the hospital for monitoring and treatment others are sent home for phototherapy. At Children's, approximately 61% of the newborns evaluated for jaundice were admitted to the hospital for further care.4

In 2004 the American Academy of Pediatrics (AAP) implemented evidence-based recommendations for the treatment of jaundice, that incorporate not only the infant's serum bilirubin concentrations but also gestational age, postnatal age, symptoms and risk factors for pathologic hyperbilirubinemia.5, 6 The AAP recommendations are the basis of all current jaundice clinical algorithms. The main treatment options according to the AAP guidelines are phototherapy, and in rare circumstances, exchange transfusions or pharmacologic treatments.2 Phototherapy is the most common treatment for jaundice and may be used in either a home-based setting or after admission to a hospital.6 Phototherapy reduces serum bilirubin levels by changing the shape and structure of bilirubin to one that is water soluble and can more simplistically be eliminated from the body through urine and stool.1 For those patients who fail phototherapy treatment or in whom the levels are exceedingly high, the use of exchange transfusions is an option within the hospital setting. Phototherapy has been successfully and safely utilized in the home-based setting to reduce the likelihood of hospital readmissions.6 Although pediatricians have successfully utilized home-based phototherapy, ED utilization of this option has been limited by access to phototherapy equipment vendors and ED provider knowledge of the criteria for outpatient management. As a result of this knowledge and access gap, the current ED care for infants with jaundice results in variation in care and over-hospitalization of infants who may be safely treated at home.

While the AAP guidelines educate physicians on the importance of evaluating infants who are 3 - 5 days of age, there is a lack of adherence to these recommendations and follow-up is often delayed. As an example, Profit et al. evaluated a large group of urban and suburban pediatricians to determine adherence with the AAP recommendations for follow-up of healthy newborn infants ≥35 weeks gestational age. Only 37% of infants in the study were seen by a pediatrician within the first 6 days of life.7 This finding is consistent with national trends that show infants frequently present to EDs when symptoms of jaundice emerge in lieu of the recommended screening.1 For example, in 2007, EDs across the United States evaluated almost 46,000 patients for neonatal jaundice. In order to reduce time to phototherapy and decrease ED length of stay8 when faced with the emergent presentation of jaundice some hospitals have implemented clinical pathways. Gomez et al. developed and implemented such a pathway through the use of a CDS tool to accurately diagnose and treat jaundice as well as to mitigate the costs that are associated with readmissions to hospitals. The authors found that the clinical pathway was useful for clarifying the decision process for clinicians by helping to educate clinicians about treatment options for jaundice them gain while highlighting inconsistencies in their routine protocols.9 Other authors have similarly reported that clinical pathways can help to reduce irregularities and discrepancies in neonatal jaundice care.10 Thus, the available literature would support that clinical pathways for neonatal jaundice can be useful and can lead to meaningful improvements in patient care.

Key strategies for improving adherence to current jaundice clinical pathways are to increase ED clinician knowledge and improve access outpatient phototherapy. An electronic, Cerner-based CDS tool, such as the one we propose, would provide clinicians with information at the point of care and would be incorporated into the ED workflow. This approach utilizes algorithms developed from evidenced based guidelines to standardize the treatment of neonatal jaundice and stratify patients into diagnostic risk groups based on particular aspects of the history, physical examination and laboratory data. The goal is to standardize the care in order to promote safe, cost-effective as well as appropriate care for all infants. This is especially important in the ED, where there is a high volume of acutely ill patients for whom management decisions must be made both accurately and quickly. This includes the rapid recognition of who is at risk of more serious complications and conditions such as kernicterus and who can safely be discharged home.3 Finally, the ordering, delivery, and set-up of home phototherapy equipment must require minimal effort by the ED clinician. We propose to leverage our electronic health record (EHR) system to streamline ordering and our well established home nursing organization to conduct home nursing visits to address these barriers to adherence with jaundice clinical pathways.

Research Question Will a clinical decision support tool for jaundice promote appropriate use of home photo therapy and reduce hospital admissions for patients at risk for jaundice?

Design This is a prospective, interrupted time series trial.

Methods We will measure resource utilization (i.e. laboratory use, hospital admission) retrospectively for 48 months pre-intervention in children identified at risk for jaundice presenting for care in a Children's Emergency Departments. We will then implement the jaundice-CDS over a 2-month period and measure resource utilization for 18 months post intervention. Rates of unplanned ED or hospital visits, use of exchange-transfusion and mortality will be monitored as safety outcomes.

Jaundice-CDS is composed of two components. The first, MD Alert, triggered at initial provider login will cognitively prime the ED provider toward use of Jaundice-CDS. The second consists of a pre-populated order-set which provides targeted recommendations and guidance on use of photo-therapy and criteria for hospital admission. Both are based on the currently accepted pediatric guideline for management of this condition.

MD ALERT:

A provider EHR-based alert will trigger for infants identified by triage who are meet eligibility criteria. This alert will serve to remind the clinician of the existence of a Jaundice order set, the availability of home nursing and home photo-therapy.

ORDER SET:

When the clinician begins the process of ordering any laboratory tests, they will be encouraged to utilize the Jaundice order-set. The order-set will contain recommendation on the most appropriate laboratory tests to obtain, criteria for admission to the hospital, as well as pre-defined orders for obtaining a home nursing referral and delivery of home photo-therapy equipment. A link will also be provided to "bilitool.org", an online resource for calculating a neonates risk for jaundice.

Analysis We will use logistic regression to assess, after controlling for relevant clinical factors, the odds of ordering a specific laboratory test (e.g., CBC, BMP, Coombs, etc.) in the group of patients seen during implementation of the CDS compared to the odds of such an order among patients arriving prior to the implementation of the CDS. Similar to the analysis of laboratory tests, we will use logistic regression to estimate odds ratios for admission and for home-based phototherapy among patients presenting to the ED with jaundice symptoms before and after the implementation of the CDS. We will use linear regression to compare total cost per encounter for all patients seen in the ED before the implementation of the CDS to total costs for patients seen in the ED post-implementation. In addition to ED costs, total costs of care will include any inpatient costs for patients admitted, and they will include costs for all lab tests. We will also compare costs pre- and post-implementation for those admitted to the hospital and for those discharged home.

ELIGIBILITY:
Inclusion Criteria:

* Patients are birth to 7 days post-natal age
* Present in Minneapolis or St Paul ED during the pre-implementation or implementation period with a chief complaint of jaundice.

Exclusion Criteria:

* Children born prematurely
* Concern for sepsis or bacterial infection
* In-born error of metabolism
* Metabolic disease
* Positive newborn screen (e.g. Sickle Cell Disease, Cystic Fibrosis)

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ED patients presenting with jaundice.
Sampling Method: Non-Probability Sample
Enrollment: 925 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Laboratory Testing Utilization | 18 months after clinical decision rule implemented
  We will use logistic regression to assess, after controlling for relevant clinical factors, the odds of ordering a specific laboratory test (e.g., CBC, BMP, Coombs, etc.) in the group of patients seen during implementation of the CDS compared to the odds of such an order among patients arriving prior to the implementation of the CDS. We will also use linear regression, controlling for relevant clinical variables, to estimate the impact of the CDS on the number of tests ordered in total for patients presenting to the ED with jaundice symptoms.
Reduced Admission/increase in home therapy utlization | 18 months after clinical decision rule implemented
  Similar to the analysis of laboratory tests, we will use logistic regression to estimate odds ratios for admission and for home-based phototherapy among patients presenting to the ED with jaundice symptoms before and after the implementation of the CDS.
Reduced Medical Expenditures | 18 months after clinical decision rule implemented
  Costs of all medical services within 2 weeks of the index ED visit will be captured from insurance claims data. Hospital-based costs for will be assessed from the Hospital charge master. While the goals of the CDS are to reduce hospital admission, the CDS may inadvertently lead to overuse of other diagnostic procedures such as lab tests or consultations. In addition, by discouraging admission, the CDS may result in prolonged observation periods in the ED or an inpatient unit. To capture all potential costs related to the treatment episode, we will include all billed medical services occurring at the ED visit and during the subsequent 14 days. This time window should include the most common complications associated with Jaundice.

CONTACTS AND LOCATIONS:
Overall Officials: Anupam B Kharbanda, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (2):
- United States (2):
  - Children's Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Hopsitals and Clinics of Minnesota, Saint Paul, Minnesota